CLINICAL TRIAL: NCT00152997
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Pramipexole With the Dose Range From 0.125 mg to 0.75 mg Orally Once Daily for 6 Weeks in Patients With Primary Restless Legs Syndrome.
Brief Title: Pramipexole (BI-Sifrol®) Orally Once Daily for 6 Weeks in Patients With Primary Restless Legs Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 248.557
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

INTERVENTIONS:
Drug: Pramipexole 0.125 mg tablets
Drug: Pramipexole 0.125 mg tablets Placebo

SUMMARY:
The objective of this trial is to investigate the efficacy and safety of pramipexole (0.125-0.75 mg) orally once daily as compared with placebo for 6 weeks in patients with primary restless legs syndrome (RLS) and to investigate the reliability of the Japanese version of the RLS rating scale by the International Restless Legs Syndrome Study Group (IRLSSG) as a sub-study.

ELIGIBILITY:
Inclusion Criteria:

According to the essential diagnostic criteria for RLS of NIH and IRLSSG, the following four all criterias must be presented:

1. An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in legs
2. The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying or sitting
3. The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues
4. The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night

   * PLM (during time in bed) index of at least 5 per hour (in the worst affected leg) at Visit 3
   * Total score of RLS severity scale-Japanese version by IRLSSG > 15 at Visit 3
   * At least 1 time per week of RLS symptoms interfering with sleep within the last one month at Visit 1.

Exclusion Criteria:

1. Pre-menopausal women who meet any one of the following (1) - (3):

   * Pregnant or possibly pregnant
   * In lactation
   * Desire to be pregnant during study period Even when a patient was confirmed not to fall under the criteria above at initiation of study, if the patient is of childbearing potential, pregnancy tests should be performed when possible. If pregnancy test is positive, the investigational product should be discontinued.
2. Males not using an adequate form of contraception.
3. Patients who took the neuroleptics within 4 weeks before the screening Visit 1, or neuroleptic-induced akathisia.
4. Patients who can not stop the treatment with medication or dietary supplements, which could significantly influence RLS symptoms to wash-out at least 14 days before drug administration (refer to Appendix 3 for prohibited medication), e.g. dopaminergic drugs (levodopa or dopamine agonists) or antidopaminergic drugs (neuroleptics or metoclopramide etc.), MAO inhibitors, sympathomimetics, antidepressants, hypnotics, any benzodiazepines, antiepileptics, opioids, clonidine, magnesium, ferrous salts, folic acid, vitamin B12, antihistaminics, lithium, melatonin.
5. Patients with diabetes mellitus requiring insulin therapy.
6. Patients with microcytic anemia at investigators discretion.
7. History or clinical signs of peripheral neuropathy (PNP) of any origin in physical, neurological examination, myelopathy or multiple sclerosis or any other neurological disease, with potential to secondarily cause RLS symptoms.
8. Other sleep disorder, such as, REM sleep behaviour disorder, narcolepsy or sleep apnea syndrome (with AHI >15 at Visit 3, or a history of loud snoring occurring at least 5 nights a week combined with a history of breathing pauses during sleep and excessive daytime sleepiness).
9. Clinically significant renal disease or creatinine higher than upper limit of normal (ULN) at screening.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-08; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Decrease in periodic limb movements during time in bed index (PLMI) in the PSG

SECONDARY OUTCOMES:
Total score of RLS severity scale-J by IRLSSG, Periodic Limb Movements during Sleep Index (PLMSI) in the PSG Periodic Limb Movements during Wakefulness Index (PLMWI) in the PSG Periodic Limb Movements in Sleep with Arousal Index (PLMAI) in the PSG )

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (7):
- Japan (7):
  - Boehringer Ingelheim Investigational Site, Akita, Akita
  - Boehringer Ingelheim Investigational Site, Kochi, Kochi
  - Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - Boehringer Ingelheim Investigational Site, Otaru,Hokkaido
  - Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - Boehringer Ingelheim Investigational Site, Shibuya,Tokyo
  - Boehringer Ingelheim Investigational Site, Takatsuki, Osaka

REFERENCES:
- [Derived] Inoue Y, Oka Y, Kagimura T, Kuroda K, Hirata K. Reliability, validity, and responsiveness of the Japanese version of International Restless Legs Syndrome Study Group rating scale for restless legs syndrome in a clinical trial setting. Psychiatry Clin Neurosci. 2013 Sep;67(6):412-9. doi: 10.1111/pcn.12074. Epub 2013 Aug 5. PMID 23910574